CLINICAL TRIAL: NCT04976686
Title: Studying the Impact of a Low Carbohydrate Diet on the Small Intestinal Microbiota
Brief Title: Low Carbohydrate Small Intestine Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted after intervention group completed. Control group with only 3 participants
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-01262
Record Dates: First submitted 2021-07-12; First posted 2021-07-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diet, Healthy
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: First phase will be purely observational, second phase involves diet modification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All study participants (Experimental): All participants will undergo sample collection during their regular diet and after modification of their diet to a low carbohydrate diet
  Interventions: Other: Diet modification

INTERVENTIONS:
Other: Diet modification — Participants will reduce their carbohydrate consumption to 80g daily

SUMMARY:
The investigators will recruit probands with a ileo- or colostoma that are otherwise in good general health and analyse the stomal fluids for their microbiota composition. Sampling will be performed over a time span of 28 days, after 14 days probands will modify their base-line diet to a low carbohydrate diet.

DETAILED DESCRIPTION:
Additionally to stoma fluids which will be analyzed for their microbiota composition the investigators will also collect skin samples to analyze for microbiota composition and urine to analyze for metabolite composition.

Low carbohydrate diet will allow for consumption of 80g complex carbohydrates per day, simple sugars will have to be avoided completely

ELIGIBILITY:
Inclusion Criteria:

* Ileostomy or colostomy
* Good general health
* Written informed consent

Exclusion Criteria:

* Major metabolic diseases that prevent adherence to low carbohydrate diet
* Participation in other clinical trial interfering with study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Assessment of microbiota profile by 16S sequencing before and after diet modification for significant differences | 28 days
  Sample content will be measured by 16S sequencing, ecological distances will be assessed by beta-diversity

SECONDARY OUTCOMES:
Relative changes of total metabolite abundance in urine | 28 days
  The whole metabolite composition will be assessed by an untargeted screen done with mass spectrometry
Analysis of microbiota metabolic potential (microbiome DNA coding for enzymes) after shotgun sequencing | 28 days
  The total DNA content of the samples will be annotated for for known metabolic active enzymes to assess functionality
Analysis of microbiota biomass | 28 days
  The samples will be analysed for the number of bacteria present in them
Changes of further metagenomic microbiome composition (viral, eucaryotic DNA) | 28 days
  The DNA of the samples will be screened for parts belonging to viruses or eucaryotic cells
Culturing of microbiota if appropriate (in vitro) | 28 days
  If of interest, culturing of specific bacterial strains will be attempted in vitro with the aim to recreate in vivo observations

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, Prof. Dr. med., Principal Investigator — University Clinic for Visceral Surgery and Medicine
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Sharing of raw sequencing data as electronic supplement to publication (e.g. by entry on database)
Time Frame: upon publication, unlimited
Access Criteria: Open access